CLINICAL TRIAL: NCT05564585
Title: Immediate Effect oF Kinesio Taping on Calf Soreness and Extensibility Among Endurance Athletes
Brief Title: Effect Kinesio Taping on Acute-onset Muscle Soreness and Calf Muscle Extensibility Among Endurance Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AMIR IQBAL (Other)
Collaborators: Hamdard University (Other)
Responsible Party: Sponsor-Investigator, AMIR IQBAL, Researcher, King Saud University
Organization: King Saud University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: JHIEC-03/18
Record Dates: First submitted 2022-09-25; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Muscle Soreness
Keywords: Kinesio tape; Sham tape; Ankle dorsiflexion; Range of motion; Pain; Muscle soreness
MeSH Terms: conditions — Myalgia; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Tape (Experimental): Kinesio Tape was applied over the Calf Muscle on Either leg.
  Interventions: Other: Kinesio Taping
- Sham Tape (Sham Comparator): Sham Tape was applied over the Calf Muscle on Either leg.
  Interventions: Other: Sham Taping

INTERVENTIONS:
Other: Kinesio Taping — Kinesio tape was applied over the calf muscle of either leg.
  Arms: Kinesio Tape
Other: Sham Taping — The sham tape was applied over the calf muscle of either leg.
  Arms: Sham Tape

SUMMARY:
In recent years, athletes have frequently utilized Kinesio tape (KT) to enhance their performance. Despite widespread use, data regarding its efficacy and mechanism of action is lacking among healthy endurance athletes. This study aims to determine the effect of KT application on acute-onset muscle soreness and the extensibility of the calf muscles in endurance athletes.

DETAILED DESCRIPTION:
The study followed a single-blinded one-arm crossover repeated-measures randomized controlled design and included fifty-five endurance athletes (mean age, 16.40±2.69) from different stadia in Delhi, India. Outcome measures, including the ankle dorsiflexion range of motion (ADFROM), were measured using a universal goniometer before, immediately after application of either KT or Sham tape, and after treadmill running. However, the pain due to acute-onset muscle soreness was measured using a numeric pain rating scale (NPRS) immediately, 10 min, and 30 min after treadmill running.

ELIGIBILITY:
Inclusion Criteria:

* Endurance athletes, including Cyclists, Badminton players, Long-distance runners
* Both males and females aged between 10-20 years
* Having BMI within the normal range (19-25)
* Cooperation in the study

Exclusion Criteria:

* Other than endurance athletes
* Aged less than Ten and more than 20 years
* BMI fall beyond the normal range, either underweight or overweight
* Musculoskeletal injuries, skin problems
* Non-cooperation in the study

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2018-11-18 (Actual); Study Completion 2019-01-20 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 1 Day
  NPRS was used to measure the level of pain. NPRS measures pain from a scale of zero to Ten where zero represent No pain and Ten represent maximum pain. Greater the score worse the pain.
Range of Motion | 1 Day
  Ankle active Dorsiflexion Range of Motion (ADFROM) was measured by a standard Goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: AMIR IQBAL, Principal Investigator — King Saud University
Locations (1):
- Rehabilitation Research Chair, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No